CLINICAL TRIAL: NCT03188666
Title: A Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Effects on Heterotopic Bone Formation of REGN2477 in Patients With Fibrodysplasia Ossificans Progressiva
Brief Title: A Study to Examine the Safety, Tolerability and Effects on Abnormal Bone Formation of REGN2477 in Patients With Fibrodysplasia Ossificans Progressiva
Acronym: LUMINA-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R2477-FOP-1623; 2016-005035-33 (EudraCT Number)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Fibrodysplasia Ossificans Progressiva
MeSH Terms: conditions — Myositis Ossificans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN2477 (Experimental)
  Interventions: Drug: REGN2477
- Placebo (Experimental)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: REGN2477 — Pharmaceutical form: liquid product for injection/infusion; Route of administration: Intravenous (IV); Administered during treatment periods 1 and 2.
  Arms: REGN2477
Drug: Matching placebo — Pharmaceutical form: Liquid product for injection/infusion; Route of administration: Intravenous (IV); Administered during treatment period 1 only.
  Arms: Placebo

SUMMARY:
This is a three period study design consisting of a 6-month, randomized, double-blind placebo-controlled treatment (period 1) followed by a 6-month, open-label treatment (period 2) and a follow-up treatment period (period 3).

Primary safety objective of the study is to assess the safety and tolerability of REGN2477 in male and female patients with fibrodysplasia ossificans progressiva (FOP).

Primary efficacy objective of the study is to assess the effect of REGN2477 versus placebo on the change from baseline in heterotopic ossification (HO) in patients with FOP, as determined by 18-NaF uptake in HO lesions by positron emission tomography (PET) and in total volume of HO lesions by computed tomography (CT).

Key Secondary objectives are:

* To compare the effect of REGN2477 versus placebo on pain due to FOP, as measured by the area under the curve (AUC) for pain based on daily pain numeric rating scale (NRS) scores
* To assess the effect of REGN2477 versus placebo on the change from baseline in HO, as determined by the number of new HO lesions identified by 18F-NaF PET or by CT
* To assess the effect of REGN2477 versus placebo on the change from baseline in 18F-NaF standardized uptake value maximum (SUVmax) of individual active HO site(s) by PET
* To assess the effect of REGN2477, between week 28 and week 56, on the number, activity, and volume of HO lesions identified by 18F-NaF PET or by CT in patients who switch from placebo to REGN2477 at week 28 versus the same patients between baseline and week 28
* To assess the effect of REGN2477 versus placebo on the change from baseline in biochemical markers of bone formation
* To characterize the concentrations of total activin A at baseline and over time following the first dose of study drug
* To characterize the concentration-time profile (pharmacokinetics [PK]) of REGN2477 in patients with FOP
* To assess the immunogenicity of REGN2477

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women 18 to 60 years of age at screening.
* Clinical diagnosis of FOP (based on findings of congenital malformation of the great toes, episodic soft tissue swelling, and/or progressive heterotopic ossification (HO)).
* Confirmation of FOP diagnosis with documentation of any ACVR1 mutation.
* FOP disease activity within 1 year of screening visit. FOP disease activity is defined as pain, swelling, stiffness, and other signs and symptoms associated with FOP flare-ups; or worsening of joint function, or radiographic progression of heterotopic ossifications (increase in site or number of HO lesions) with/without being associated with flare-up episodes.
* Willing and able to undergo PET and CT imaging procedures and other procedures as defined in this study.

Key Exclusion Criteria:

* Significant concomitant illness or history of significant illness such as, but not limited to cardiac, renal, rheumatologic, neurologic, psychiatric, endocrine, metabolic or lymphatic disease, that in the opinion of the study investigator might confound the results of the study or pose additional risk to the patient by their participation in the study.
* Previous history or diagnosis of cancer.
* Use of bisphosphonate within 1 year of screening.
* Concurrent participation in another interventional clinical study, or a non-interventional study with radiographic measures or invasive procedures (e.g. collection of blood or tissue samples). Participation in the FOP Connection Registry or other studies in which participants complete study questionnaires are allowed.
* Treatment with another investigational drug, denosumab, imatinib or isotretinoin in the last 30 days or within 5 half-lives of the investigational drug, whichever is longer.
* Pregnant or breastfeeding women.
* Male and women of childbearing potential participants who are unwilling to practice highly effective contraception.

Note: Other protocol defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (11):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Toronto General Hospital, Toronto, Ontario, Canada
- France (2):
  - Hopital Cochin, Paris
  - Hopital Lariboisiere,Hospitalier Universitaire Nord, Paris
- Giannina Gaslini Institute, Genova, Italy
- VU University Medical Center, Amsterdam, North Holland, Netherlands
- Szpital Wojewodzki Nr 2, Rzeszów, Poland
- Hospital Universitario Ramon y Cajal, Madrid, Spain
- Royal National Orthopaedic Hospital, Brockley Hill, Stanmore, Middlesex, United Kingdom

REFERENCES:
- [Derived] de Ruiter RD, Botman E, Teunissen BP, Lammertsma AA, Boellaard R, Raijmakers PG, Schwarte LA, Nieuwenhuijzen JA, Gonzalez Trotter D, Eekhoff EMW, Yaqub M. Performance of simplified methods for quantification of [18F]NaF uptake in fibrodysplasia ossificans progressiva. Front Nucl Med. 2024 Jul 22;4:1406947. doi: 10.3389/fnume.2024.1406947. eCollection 2024. PMID 39381032
- [Derived] Di Rocco M, Forleo-Neto E, Pignolo RJ, Keen R, Orcel P, Funck-Brentano T, Roux C, Kolta S, Madeo A, Bubbear JS, Tabarkiewicz J, Szczepanek M, Bachiller-Corral J, Cheung AM, Dahir KM, Botman E, Raijmakers PG, Al Mukaddam M, Tile L, Portal-Celhay C, Sarkar N, Hou P, Musser BJ, Boyapati A, Mohammadi K, Mellis SJ, Rankin AJ, Economides AN, Trotter DG, Herman GA, O'Meara SJ, DelGizzi R, Weinreich DM, Yancopoulos GD, Eekhoff EMW, Kaplan FS. Garetosmab in fibrodysplasia ossificans progressiva: a randomized, double-blind, placebo-controlled phase 2 trial. Nat Med. 2023 Oct;29(10):2615-2624. doi: 10.1038/s41591-023-02561-8. Epub 2023 Sep 28. PMID 37770652
- [Derived] Vanhoutte F, Liang S, Ruddy M, Zhao A, Drewery T, Wang Y, DelGizzi R, Forleo-Neto E, Rajadhyaksha M, Herman G, Davis JD. Pharmacokinetics and Pharmacodynamics of Garetosmab (Anti-Activin A): Results From a First-in-Human Phase 1 Study. J Clin Pharmacol. 2020 Nov;60(11):1424-1431. doi: 10.1002/jcph.1638. Epub 2020 Jun 18. PMID 32557665
- [Derived] Aykul S, Corpina RA, Goebel EJ, Cunanan CJ, Dimitriou A, Kim HJ, Zhang Q, Rafique A, Leidich R, Wang X, McClain J, Jimenez J, Nannuru KC, Rothman NJ, Lees-Shepard JB, Martinez-Hackert E, Murphy AJ, Thompson TB, Economides AN, Idone V. Activin A forms a non-signaling complex with ACVR1 and type II Activin/BMP receptors via its finger 2 tip loop. Elife. 2020 Jun 9;9:e54582. doi: 10.7554/eLife.54582. PMID 32515349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 participants were screened, out of which, 44 participants were randomized and treated.
Pre-assignment Details: This was a three period study design which consisted of a 6-month (28 weeks), randomized, double-blind placebo-controlled treatment period (Period 1) followed by a 6-month (28 weeks), open-label treatment period (Period 2) and a 20 week follow-up treatment period (Period 3). Participants could continue receiving REGN2477 every 4 weeks beyond week 76 provided that no safety signals were identified.
Groups:
- Placebo: Participants received a single dose of placebo matched to REGN2477 intravenous (IV) infusion every 4 weeks (Q4W) for up to 28 weeks during Period 1.
- REGN2477 10 mg/kg Q4W: Participants received a single dose of REGN2477 10 milligrams per kilogram (mg/kg) IV infusion every 4 weeks (Q4W) for up to 28 weeks during Period 1.
- Placebo/REGN2477 10 mg/kg Q4W: Participants who were in the placebo group in Period 1 crossed over to receive a single dose of REGN2477 IV infusion Q4W for 28 weeks during Period 2 followed by 20 weeks during Period 3.
- REGN2477/REGN2477 10 mg/kg Q4W: Participants who were in the REGN2477 group in Period 1 continued treatment with a single dose of REGN2477 IV infusion Q4W for additional 28 weeks during Period 2 followed by 20 weeks during Period 3.
Period: Period 1 (28 Weeks Double-blind)
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Started | 24 | 20 | 0 | 0
Completed | 24 | 19 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 2 (28 Weeks Open-label)
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Started | 0 | 0 | 24 | 19
Completed | 0 | 0 | 24 | 18
Not Completed | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1
Period: Period 3 (20 Weeks Follow-up)
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Started | 0 | 0 | 24 | 18
Completed | 0 | 0 | 21 | 16
Not Completed | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants and was based on the treatment allocated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W | Total
Number analyzed (Participants) | 24 | 20 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (8.54) | 27.3 (8.67) | 27.6 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 22 | 17 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Total Lesion Activity by fluorine-18 sodium fluoride (18 F-NaF) PET (AHO Analysis Set) [Mean (Standard Deviation); unit: gram (g)] — 18^F-NaF positron emission tomography (PET) imaging was used to assess lesion and disease activity. Population: The baseline-active HO analysis set (AHO) includes all randomized patients who had at least one active HO lesion at baseline; it is based on the treatment allocated (as randomized).
  gram (g) | 473.40 (348.373) | 418.18 (372.801) | 448.30 (356.510)
Total Volume of HO Lesions as Assessed by Computed Tomography (CT) (AHO Analysis Set) [Mean (Standard Deviation); unit: cubic centimeter (cm^3)] — CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. The baseline-Active Heterotopic ossification (AHO) analysis set includes all randomized patients who had at least one active HO lesion at baseline; it is based on the treatment allocated (as randomized).
  cubic centimeter (cm^3) | 235.78 (253.329) | 251.43 (327.881) | 242.89 (286.167)
Total Lesion Activity by 18F-NaF PET (AHOC Analysis Set) [Mean (Standard Deviation); unit: gram (g)] — 18^F-NaF positron emission tomography (PET) imaging was used to assess lesion and disease activity. Population: The baseline-active HO classic ACVR1 [R206H] mutation analysis set (AHOC) includes all randomized patients with the classic ACVR1 [R206H] mutation and who had at least one active HO lesion(s) at baseline, as defined by 18F-NaF PET positivity; it is based on the treatment allocated (as randomized)
  gram (g)
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 464.27 (350.479) | 418.18 (372.801) | 442.32 (357.581)
Total Volume of HO Lesions as Assessed by CT (AHOC Analysis Set) [Mean (Standard Deviation); unit: cubic centimeter (cm^3)] — CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Population: The baseline-active HO classic ACVR1 [R206H] mutation analysis set (AHOC) includes all randomized patients with the classic ACVR1 [R206H] mutation and who had at least one active HO lesion(s) at baseline, as defined by 18F-NaF PET positivity; it is based on the treatment allocated (as randomized)
  cubic centimeter (cm^3)
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 239.72 (263.813) | 251.43 (327.881) | 245.29 (292.408)
Fibrodysplasia Ossificans Progressiva (FOP) Genetic Mutation [Count of Participants; unit: Participants]
  Active HO classic ACVR1 (R206H) | 22 | 20 | 42
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Treatment-emergent adverse events (TEAEs) are adverse events not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period. A serious TEAE was defined as any untoward medical occurrence that resulted in any of following outcomes not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. Number of participants with TEAEs and Serious TEAEs are reported.
Time Frame: Up to Week 28
Population: The safety analysis set included all randomized participants who received any study drug and was analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
Participants
  Participants with at least one TEAE | 24 | 20
  Participants with at least one serious TEAE | 2 | 4

2. Primary Outcome: Period 1: Number of Participants With TEAEs by Severity
Description: Severity of TEAEs were graded as follows: Mild: Does not interfere in a significant manner with the participant's normal functioning level. It may be an annoyance. Prescription drugs are not ordinarily needed for relief of symptoms but may be given because of personality of the participants. Moderate: Produces some impairment of functioning but is not hazardous to health. It was uncomfortable or an embarrassment. Treatment for symptom may be needed. Severe: Produces significant impairment of functioning or incapacitation and was a definite hazard to the participant's health. Treatment for symptom may be given and/or participants hospitalized. Number of participants with TEAEs by severity is reported.
Time Frame: Up to Week 28
Population: The safety analysis set included all randomized participants who received any study drug and was analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
Participants
  Participants with at least one Mild TEAE | 9 | 7
  Participants with at least one Moderate TEAE | 12 | 10
  Participants with at least one Severe TEAE | 3 | 3

3. Primary Outcome: Period 1: Time-Weighted Average (Standardized Area Under the Curve [AUC]) of the Percent Change From Baseline in Total Lesion Activity by Fluorine-18-labeled Sodium Fluoride (18^F-NaF) Positron Emission Tomography (PET) at Week 28 (AHO)
Description: 18^F-NaF PET is used to assess lesion and disease activity. Time-weighted average (standardized area under the curve [AUC]) of the percent change from baseline in total lesion activity by 18^F-NaF PET up to Week 28 in AHO analysis set is reported.
Time Frame: Baseline and Week 28
Population: Baseline-active heterotopic ossification analysis set (AHO) included all randomized participants who had at least one active HO lesion at baseline; and was based on the treatment allocated (as randomized).
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
Percent Change | 16.6 (9.11) | -8.1 (9.93)
Statistical Analysis 1: Comparison: Placebo vs REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.0741, ANCOVA; Least Square Mean Difference = -24.6, 95% CI 2-sided [-51.8 to 2.5]

4. Primary Outcome: Period 1: Percent Change From Baseline in the Total Volume of HO Lesions as Assessed by Computed Tomography (CT) at Week 28 (AHO)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Percent change from baseline in the total volume of HO lesions as assessed by CT during Period 1 at Week 28 is reported.
Time Frame: Week 28
Population: AHO analysis set included all randomized participants who had at least one active HO lesion at baseline was based on the treatment allocated (as randomized).
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
Percent Change | 32.0 (18.66) | 7.1 (20.43)
Statistical Analysis 1: Comparison: Placebo vs REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.3726, Mixed Model with Repeated Measure (MMRM); Least Square Mean Difference = -24.9, 95% CI 2-sided [-80.8 to 30.9]

5. Primary Outcome: Period 2: Number of New HO Lesions as Assessed by CT at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. HO detectable by CT that developed after baseline are referred to as "new HO lesions." Number of new HO lesions as assessed by CT at Week 56 relative to Week 28 scan is reported.
Time Frame: Week 28, Week 56
Population: COVID-19 mITT: All AHO participants who received a treatment in Period 2 for whom at least 1 post-Week 28 scan was collected and the period between any consecutive doses was less than 9 weeks (63 days) before the 1st post-week 28 scan. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure. Separate analyses were conducted from week 56 relative to baseline for participants on treatment during both periods (REGN2477/REGN2477) as planned.
Measure: Number; unit: New HO Lesions
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
New HO Lesions | 0
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W; Compared number of new lesions per participant by CT at week 28 (relative to baseline) and week 56 (relative to week 28); Test type: Superiority; p = 0.0039, Wilcoxon signed rank test — Week 56 vs. Week 28

6. Primary Outcome: Period 1: Time-weighted Average (Standardized AUC) of the Percent Change From Baseline in Total Lesion Activity Assessed by 18^F-NaF PET at Week 28 (AHOC)
Description: 18^F-NaF PET is used to assess lesion and disease activity. Time-weighted average (Standardized AUC) of the percent change from baseline in total lesion activity as assessed by 18^F-NaF PET in Active HO Classic ACVR1 Mutation (AHOC) analysis set up to Week 28 is reported.
Time Frame: Week 28
Population: AHOC analysis set included all randomized participants with the classic ACVR1 [R206H] mutation and who had at least one AHO at baseline, as defined by 18^F-NaF PET positivity; and was based on the treatment allocated (as randomized). "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22 | 20
Percent Change | 17.6 (9.73) | -8.0 (10.14)
Statistical Analysis 1: Comparison: Placebo vs REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.0756, ANCOVA; Least Square Mean Difference = -25.6, 95% CI 2-sided [-53.9 to 2.8]

7. Primary Outcome: Period 1: Percent Change From Baseline in the Total Volume of HO Lesions as Assessed by CT at Week 28 (AHOC)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Percent change from baseline in the total volume of HO lesions was assessed by CT at Week 28 in AHOC analysis set is reported.
Time Frame: Week 28
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22 | 20
Percent Change | 34.9 (19.90) | 7.0 (20.87)
Statistical Analysis 1: Comparison: Placebo vs REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.3407, Mixed Model with Repeated Measure (MMRM); Least Square Mean Difference = -27.8, 95% CI 2-sided [-86.1 to 30.5]

8. Secondary Outcome: Period 1: Time-weighted Average (Standardized AUC) of the Change From Baseline in Daily Pain Due to Fibrodysplasia Ossificans Progressiva (FOP) Assessed by Daily Numeric Rating Scale (NRS) at Week 28 (AHO)
Description: The pain NRS is a patient reported outcome (PRO) used by participants to rate their pain associated with FOP. Participants were asked to rate their pain on a scale that ranges from "0" (no pain) to "10" (worst possible pain), where the highest score indicated worst outcome. Time-weighted average (Standardized AUC) of the change from baseline in daily pain due to FOP assessed by daily NRS at Week 28 in AHO analysis set is reported.
Time Frame: Week 28
Population: AHO analysis set included all randomized participants who had at least one active HO lesion at baseline; based on the treatment allocated (as randomized). "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 23 | 18
Score on a Scale | -0.17 (0.205) | -0.51 (0.231)
Statistical Analysis 1: Comparison: Placebo vs REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.2656, ANCOVA; Least Square Mean Difference = -0.34, 95% CI 2-sided [-0.96 to 0.27]

9. Secondary Outcome: Period 1: Time-weighted Average (Standardized AUC) of the Change From Baseline in Daily Pain Due to FOP, Assessed by Daily NRS at Week 28 (AHOC)
Description: The pain NRS is a PRO used by participants to rate their pain associated with FOP. Participants were asked to rate their pain on a scale that ranges from "0" (no pain) to "10" (worst possible pain), where the highest score indicated worst outcome. Time-Weighted average (standardized AUC) of the change from baseline in daily pain due to FOP assessed by daily NRS at Week 28 in AHOC analysis set is reported.
Time Frame: Week 28
Population: as for outcome 6
Measure: Least Squares Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 21 | 18
Score on a Scale | -0.12 (0.221) | -0.48 (0.237)
Statistical Analysis 1: Comparison: Placebo vs REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.2651, ANCOVA; Least Square Mean Difference = -0.36, 95% CI 2-sided [-1.01 to 0.29]

10. Secondary Outcome: Period 1: Percent Change From Baseline in 18^F-NaF SUVmax of Individual Active HO Site(s) Assessed by 18^F-NaF PET at Week 8 (AHOC)
Description: Standardized uptake value max (SUVmax) was a measurement of the maximum radiopharmaceutical uptake within the volume of interest. Relative accuracy of a particular radiotracer in a particular tissue is determined by expressing the absolute accuracy (obtained in the primary outcome measure) in terms of percent difference between SUVmax values obtained from PET/CT. Percent Change in 18^F-NaF SUVmax of Individual Active HO Site(s) assessed by 18^F-NaF PET in AHOC analysis set is reported.
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22 | 20
Percent Change | -6.7 (28.79) | -21.6 (30.25)

11. Secondary Outcome: Period 1: Percent Change From Baseline in 18^F-NaF SUVmax of Individual Active HO Site(s) as Assessed by 18^F-NaFPET at Week 8 (AHO)
Description: Percent change in 18^F-NaF SUVmax of individual active HO site(s) as assessed by 18^F-NaF PET at Week 8 in AHO analysis set is reported.
Time Frame: Week 8
Population: AHO analysis set included all randomized participants who had at least one active HO lesion at baseline; based on the treatment allocated (as randomized).
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
Percent Change | -7.9 (28.80) | -21.6 (30.25)

12. Secondary Outcome: Period 1: Change From Baseline in Number of HO Lesions as Assessed by 18^F-NaF PET at Week 28 (AHOC)
Description: Change from baseline in number of HO lesions was assessed by 18^F-NaF PET at Week 28 in AHOC analysis set is reported.
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: HO Lesions
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22 | 20
HO Lesions | -1.0 (2.66) | -2.3 (2.24)

13. Secondary Outcome: Period 1: Change From Baseline in Number of HO Lesions as Assessed by 18^F-NaF PET at Week 28 (AHO)
Description: Change from baseline in number of HO lesions was assessed by 18^F-NaF PET in AHO analysis set is reported.
Time Frame: Week 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: HO Lesions
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
HO Lesions | -1.0 (2.59) | -2.3 (2.24)

14. Secondary Outcome: Period 1: Change From Baseline in Number of HO Lesions Detectable by CT at Week 28 (AHOC)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Change from baseline in number of HO lesions was detectable by CT using AHOC analysis set is reported.
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: HO Lesions
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22 | 20
HO Lesions | 1.2 (2.00) | -0.3 (1.34)

15. Secondary Outcome: Period 1: Change From Baseline in Number of HO Lesions Detectable by CT at Week 28 (AHO)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Change from baseline in number of HO lesions detectable by CT at Week 28 in AHO analysis set is reported.
Time Frame: Week 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: HO Lesions
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
HO Lesions | 1.2 (1.93) | -0.3 (1.34)

16. Secondary Outcome: Period 2: Number of New HO Lesions as Assessed by 18^F-NaF PET at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: Number of new HO lesions as assessed by 18^F-NaF PET at Week 56 Relative to Week 28 Scan is reported.
Time Frame: Week 28, Week 56
Population: as for outcome 5
Measure: Number; unit: New HO lesions
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
New HO lesions | 1
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W; Compared number of new lesions per participant by PET at week 28 (relative to baseline) and week 56 (relative to week 28); Test type: Superiority; p = 0.0039, Wilcoxon signed rank test — Week 56 vs. Week 28

17. Secondary Outcome: Period 2: Percentage of Participants With New HO Lesions as Assessed by CT at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Percentage of participants with new HO lesions as assessed by CT at week 56 relative to week 28 scan is reported.
Time Frame: Week 28, Week 56
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
Percentage of Participants | 0.0
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W; Compared percent of participants with new lesions by CT at week 28 (relative to baseline) and week 56 (relative to week 28); Test type: Superiority; p = 0.0027, McNemar — Week 56 vs. Week 28

18. Secondary Outcome: Period 2: Percentage of Participants With New HO Lesions as Assessed by 18^F-NaF PET at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: 18^F-NaF PET is used to assess lesion and disease activity. Percentage of participants with new HO lesions as assessed by 18^F-NaF PET at week 56 relative to week 28 scan is reported.
Time Frame: Week 28, Week 56
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
Percentage of Participants | 4.5
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W; Compared percent of participants with new lesions by PET at week 28 (relative to baseline) and week 56 (relative to week 28); Test type: Superiority; p = 0.0047, McNemar — Week 56 vs. Week 28

19. Secondary Outcome: Period 2: Number of New HO Lesions as Assessed by CT Only at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT Only: Computed Tomography (CT) assessment without reference to positron-emission tomography (PET). Number of new HO lesions as assessed by CT only at week 56 relative to week 28 scan is reported.
Time Frame: Week 28, Week 56
Population: as for outcome 5
Measure: Number; unit: New HO lesions
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
New HO lesions | 3

20. Secondary Outcome: Period 2: Percentage of Participants With New HO Lesions as Assessed by CT Only at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT Only: Computed Tomography (CT) assessment without reference to Positron-Emission Tomography (PET). Percentage of participants with new HO lesions as assessed by CT only at week 56 relative to week 28 scan is reported.
Time Frame: Week 28, Week 56
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
Percentage of Participants | 9.1

21. Secondary Outcome: Period 2 vs. Period 1: Change From Week 28 in Number of Active HO Lesions as Assessed by 18^F-NaF PET to Week 56 (Period 2) Versus the Same Participants Between Baseline and Week 28 (Period 1) (AHO COVID-19 mITT)
Description: 18^F-NaF PET is used to assess lesion and disease activity. Difference of Change from Week 28 to Week 56 as assessed by 18^F-NaF PET versus from Baseline to Week 28
Time Frame: Week 28, Week 56
Population: COVID-19 mITT: All AHO participants who received a treatment in period 2 for whom at least 1 post-Week 28 scan was collected and the period between any consecutive doses was less than 9 weeks (63 days) before the 1st post-week 28 scan. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Active lesions
Groups:
- REGN2477/REGN2477 10 mg/kg Q4W: Participants who were in the REGN2477 group in Period 1 continued treatment with a single dose of REGN2477 IV infusion Q4W for additional 28 weeks (up to Week 56) during Period 2.
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 19 | 17
Active lesions | -1.2 (4.31) | 1.3 (3.26)
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W vs REGN2477/REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.3663, Wilcoxon signed rank test — Period 2 vs. Period 1

22. Secondary Outcome: Period 2 vs. Period 1: Change From Week 28 in Number of Active HO Lesions as Assessed by CT Scan at Week 56 (Period 2) Versus the Same Participants Between Baseline and Week 28 (Period 1) (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Difference of Change from Week 28 to Week 56 as assessed by CT Scan versus from Baseline to Week 28 is reported
Time Frame: Week 28, Week 56
Population: COVID-19 mITT: All AHO participants who received a treatment in period 2 for whom at least 1 post-Week 28 scan is collected and the period between any consecutive doses was less than 9 weeks (63 days) before the 1st post-week 28 scan. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Active lesions
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22 | 18
Active lesions | -1.3 (2.40) | 0.3 (1.24)
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W vs REGN2477/REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.0010, Wilcoxon signed rank test — Period 2 vs. Period 1

23. Secondary Outcome: Period 2: Number of New HO Lesions as Assessed by CT at Week 56 Relative to Baseline (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Number of new HO lesions as assessed by CT at week 56 relative to baseline.
Time Frame: Baseline, Week 56
Population: COVID-19 mITT: All AHO participants who received a treatment in period 2 for whom at least 1 post-Week 28 scan was collected and the period between any consecutive doses was less than 9 weeks (63 days) before the 1st post-week 28 scan. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure. Separate analyses were conducted from week 56 relative to week 28 for participants on treatment during period 2 only (Placebo/REGN2477) as planned.
Measure: Number; unit: New HO Lesions
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 18
New HO Lesions | 2

24. Secondary Outcome: Period 2: Number of New HO Lesions as Assessed by CT Only at Week 56 Relative to Baseline (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT Only: Computed Tomography (CT) assessment without reference to Positron-Emission Tomography (PET); Number of new HO lesions as assessed by CT only at week 56 relative baseline is reported.
Time Frame: Week 56
Population: COVID-19 mITT: All AHO participants who receive a treatment in Period 2 for whom at least 1 post-Week 28 scan is collected and the period between any consecutive doses is less than 9 weeks (63 days) before the 1st post-week 28 scan. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure. Separate analyses were conducted from week 56 relative to week 28 for participants on treatment during period 2 (Placebo/REGN2477) as planned.
Measure: Number; unit: New HO Lesions
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 18
New HO Lesions | 1

25. Secondary Outcome: Period 2: Percentage of Participants With New HO Lesions as Assessed by CT at Week 56 Relative to Baseline (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Percentage of participants with new HO lesions as assessed by CT at week 56 relative to baseline were reported.
Time Frame: Week 56
Population: COVID-19 mITT: All AHO participants who received a treatment in Period 2 for whom at least 1 post-Week 28 scan was collected and the period between any consecutive doses was less than 9 weeks (63 days) before the 1st post-week 28 scan. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure. Separate analyses were conducted from week 56 relative to week 28 for participants on treatment during period 2 (Placebo/REGN2477) as planned.
Measure: Number; unit: Percentage of Participants
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 18
Percentage of Participants | 11.1

26. Secondary Outcome: Period 2: Number of New HO Lesions as Assessed by 18^F-NAF PET at Week 56 Relative to Baseline (AHO COVID-19 mITT)
Description: 18^F-NaF PET is used to assess lesion and disease activity. Number of new HO lesions as assessed by 18^F-NAF PET at week 56 relative to baseline is reported.
Time Frame: Week 56
Population: as for outcome 25
Measure: Number; unit: New HO Lesions
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 18
New HO Lesions | 1

27. Secondary Outcome: Period 2: Percentage of Participants With New HO Lesions as Assessed by 18^F-NaF PET at Week 56 Relative to Baseline (AHO COVID-19 mITT)
Description: 18^F-NaF PET is used to assess lesion and disease activity. Percentage of participants with new HO lesions as assessed by 18^F-NaF PET at week 56 relative to baseline.
Time Frame: Week 56
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 18
Percentage of Participants | 5.6

28. Secondary Outcome: Period 2: Total Volume of New HO Lesions as Assessed by CT at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Total volume of new HO lesions as assessed by CT at Week 56 relative to Week 28 scan.
Time Frame: Week 28, Week 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cubic centimeter (cm^3)
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
cubic centimeter (cm^3) | 0.0 (0.21)
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W; Compared total new lesion volume per participant by CT at week 28 (relative to baseline) and week 56 (relative to week 28); Test type: Superiority; p = 0.0039, Wilcoxon signed rank test — Week 56 vs. Week 28

29. Secondary Outcome: Period 2: Total Lesion Activity (TLA) Assessed by 18^F-NaF PET in New HO Lesions at Week 56 Relative to Week 28 Scan (AHO COVID-19 mITT)
Description: TLA is a measure of participant-level cumulative burden of metabolically active HO. Activity of individual HO lesions was calculated as the product of mean standard uptake value (SUVmean) and the PET volume of the active HO lesion. TLA was derived for each participant at each time point as the sum of HO lesion activity of individual target and new active HO lesions.
Time Frame: Week 28, Week 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
gram (g) | 13.2 (61.89)
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W; Compared total lesion activity per participant in new lesions by PET at week 28 (relative to baseline) and week 56 (relative to week 28); Test type: Superiority; p = 0.0273, Wilcoxon signed rank test — Week 56 vs. Week 28

30. Secondary Outcome: Period 2 vs. Period 1: Percent Change From Week 28 in TLA as Assessed by 18^F-NaF PET to Week 56 (Period 2) Versus the Same Participants Between Baseline and Week 28 (Period 1) (AHO COVID-19 mITT)
Description: Difference of Percent Change from Week 28 to Week 56 versus from Baseline to Week 28 is reported
Time Frame: Week 28, Week 56
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 21 | 17
Percent Change | -66.9 (181.06) | 14.0 (41.17)
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W vs REGN2477/REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.2123, Wilcoxon signed rank test — Period 2 vs. Period 1

31. Secondary Outcome: Period 2 vs. Period 1: Percent Change From Week 28 in the Total Volume of HO Lesions as Assessed by CT to Week 56 (Period 2) Versus the Same Participants Between Baseline and Week 28 (Period 1) (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Difference of Percent Change from Week 28 to Week 56 versus from Baseline to Week 28 is reported.
Time Frame: Week 28, Week 56
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22 | 18
Percent Change | -31.8 (132.47) | -11.1 (24.07)
Statistical Analysis 1: Comparison: Placebo/REGN2477 10 mg/kg Q4W vs REGN2477/REGN2477 10 mg/kg Q4W; Test type: Superiority; p = 0.1528, Wilcoxon signed rank test — Period 2 vs. Period 1

32. Secondary Outcome: Period 2: TLA in New HO Lesions as Assessed by 18^F-NaF PET at Week 56 Relative to Baseline (AHO COVID-19 mITT)
Description: Total Lesion Activity (TLA) is a measure of participant-level cumulative burden of metabolically active HO. TLA in New (Relative to Baseline) Lesions at Week 56 is reported.
Time Frame: Week 56
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: gram (g)
Groups:
- REGN2477/ REGN2477: Participants who were in the REGN2477 group in Period 1 continued treatment with a single-dose of REGN2477 IV infusion Q4W for additional 28 weeks (up to week 56) during Period 2.
Arm/Group | REGN2477/ REGN2477
Number analyzed (Participants) | 18
gram (g) | 0.7 (2.13)

33. Secondary Outcome: Period 2: Total Volume of New HO Lesions as Assessed by CT Only at Week 56 Relative to Baseline (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT Only: Computed Tomography (CT) assessment without reference to Positron-Emission Tomography (PET); Total volume of new HO lesions as assessed by CT only at week 56 relative to baseline is reported.
Time Frame: Week 56
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: cubic centimeter (cm^3)
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 18
cubic centimeter (cm^3) | 0.0 (0.02)

34. Secondary Outcome: Period 2: Percent Change From Baseline in TLA as Assessed by 18^F-NaF PET to Week 56 (AHO COVID-19 mITT)
Description: Percent change from baseline in TLA as assessed by 18^F-NaF PET to week 56 were reported.
Time Frame: Week 56
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 17
Percent Change | -16.4 (53.10)

35. Secondary Outcome: Period 2: Percent Change From Baseline in the Total Volume of HO Lesions as Assessed by CT to Week 56 (AHO COVID-19 mITT)
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue, and blood vessels. CT scan acquired contemporaneously to the PET scan. Percent change from baseline in the total volume of HO lesions as assessed by CT to Week 56 were reported.
Time Frame: Week 56
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 18
Percent Change | 2.6 (10.18)

36. Secondary Outcome: Period 2: Percent Change From Week 28 in SUVmax as Assessed by 18^F-NaF to Week 56 (AHO COVID-19 mITT)
Description: Percent Change from Week 28 to Week 56 is reported.
Time Frame: Week 28 to Week 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 21
Percent Change | -30.3 (15.03)

37. Secondary Outcome: Period 2: Percent Change From Baseline in 18^F-NaF PET SUVmax to Week 56 (AHO COVID-19 mITT)
Description: Percent change from baseline in 18^F-NaF PET SUVmax to week 56
Time Frame: Baseline, Week 56
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 17
Percent Change | -41.9 (29.16)

38. Secondary Outcome: Period 2: Daily Average Pain Due to FOP Measured Using the Daily NRS
Description: The pain NRS is a patient reported outcome used by participants to rate their pain associated with FOP. Participants were asked to rate their pain on a scale that ranges from "0" (no pain) to "10" (worst possible pain), where the highest score indicated worst outcome.
Time Frame: Week 28 up to Week 56
Population: COVID-19 mITT: All AHO participants who received a treatment in Period 2 for whom at least 1 post-Week 28 scan was collected and the period between any consecutive doses was less than 9 weeks (63 days) before the 1st post-week 28 scan. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure. Data were planned to be collected and analyzed only for participants switching to REGN2477 in period 2 for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
Score on a Scale | 1.60 (1.969)

39. Secondary Outcome: Period 2: Percentage of Participants With Flare-ups Assessed by Participant E-diary
Description: Percentage of participants with flare-ups starting between week 28 and week 56 as assessed by participant E-diary is reported.
Time Frame: Week 28 to Week 56
Population: COVID-19 mITT: All AHO participants who received a treatment in Period 2 for whom at least 1 post-Week 28 scan was collected and the period between any consecutive doses was less than 9 weeks (63 days) before the 1st post-week 28 scan. Data were planned to be collected and analyzed only for participants switching to REGN2477 in period 2 for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
Percentage of Participants | 13.6

40. Secondary Outcome: Period 2: Percentage of Participants With Investigator-assessed Flare-ups
Description: Percentage of participants with investigator-assessed flare-ups were reported.
Time Frame: Week 28 to Week 56
Population: as for outcome 39
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 22
Percentage of Participants | 13.6

41. Secondary Outcome: Periods 1, 2, and 3: Concentration of Total Activin A in Serum
Description: Concentration of total activin A in serum over time is reported.
Time Frame: Week 28, Week 56, Week 76
Population: The PK analysis set included all treated participants who received any study drug and who had at least 1 non-missing drug concentration following the first dose of study drug. ("Number Analyzed" equals number of participants evaluable at that time point)
Measure: Mean (Standard Deviation); unit: milligram per Liter (mg/L)
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
milligram per Liter (mg/L)
  Week 28: number analyzed (Participants) | 24 | 18
  Week 28 | 0.0000813 (0.000164) | 0.0537 (0.0116)
  Week 56: number analyzed (Participants) | 20 | 16
  Week 56 | 0.0563 (0.0172) | 0.0503 (0.0113)
  Week 76: number analyzed (Participants) | 15 | 11
  Week 76 | 0.0487 (0.0192) | 0.0497 (0.0176)

42. Secondary Outcome: Periods 1, 2, and 3: Concentrations of Functional REGN2477 in Serum
Description: Concentrations of REGN2477 capable of target binding were measured (functional drug).
Time Frame: Week 28, Week 56, Week 76
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- REGN2477 10 mg/kg Q4W: Participants who were in the REGN2477 group in Period 1 continued treatment with a single dose of REGN2477 IV infusion Q4W for additional 28 weeks (up to Week 56) during Period 2.
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W | REGN2477 10 mg/kg Q4W
Number analyzed (Participants) | 24 | 20
mg/L
  Week 28: number analyzed (Participants) | 24 | 18
  Week 28 | 0 (0) | 130 (46.6)
  Week 56: number analyzed (Participants) | 20 | 16
  Week 56 | 100 (27.3) | 122 (54.8)
  Week 76: number analyzed (Participants) | 15 | 11
  Week 76 | 113 (27.0) | 113 (23.0)

43. Secondary Outcome: Periods 1, 2, and 3: Number of Participants With Clinical Impact of Treatment-Emergent Anti-drug Antibodies (ADA) to REGN2477
Description: Immunogenicity was characterized by ADA responses & titers. Responses categories: Negative - ADA negative response at all time points, regardless of missing samples; Pre-existing immunoreactivity - ADA positive response at baseline with all post first dose negative results or positive response at baseline with all post first dose ADA responses < 9-fold over baseline titer levels; Treatment-boosted response - positive response in the assay post first dose, >= 9-fold over baseline titer levels, when baseline results are positive; Treatment-emergent response - ADA positive response in the REGN2477 ADA assay post first dose when baseline results = negative or missing.
Time Frame: Up to Week 76
Population: The Anti-Drug Antibody (ADA) analysis set included all participants who received study drug and had at least 1 non-missing ADA result following the first study dose. "Overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/ REGN2477
Number analyzed (Participants) | 24 | 19
Participants
  Negative | 24 | 18
  Pre-existing Immunoreactivity | 0 | 0
  Treatment-Boosted Response | 0 | 0
  Treatment-Emergent Response | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of study
Groups:
- REGN2477/REGN2477 10 mg/kg Q4W: Participants who were in the REGN2477 group in Period 1 continued treatment with a single dose of REGN2477 IV infusion Q4W for additional 28 weeks during Period 2 followed by 20 weeks during Period 3. Participants could continue receiving REGN2477 every 4 weeks beyond week 76 provided that no safety signals were identified.
Arm/Group | Placebo | REGN2477 10 mg/kg Q4W | Placebo/REGN2477 10 mg/kg Q4W | REGN2477/REGN2477 10 mg/kg Q4W
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/20 | 2/24 | 3/19
Serious Adverse Events (participants affected / at risk) | 2/24 | 4/20 | 6/24 | 7/19
Other Adverse Events (participants affected / at risk) | 24/24 | 20/20 | 24/24 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | REGN2477 10 mg/kg Q4W (N=20) | Placebo/REGN2477 10 mg/kg Q4W (N=24) | REGN2477/REGN2477 10 mg/kg Q4W (N=19)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | REGN2477 10 mg/kg Q4W (N=20) | Placebo/REGN2477 10 mg/kg Q4W (N=24) | REGN2477/REGN2477 10 mg/kg Q4W (N=19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 7 (8) | 8 (16) | 9 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (19) | 5 (6) | 6 (18) | 8 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (4) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (5) | 2 (2) | 4 (13)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 7 (9) | 6 (13)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 1 (3) | 4 (10)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calcification of muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (14) | 10 (28) | 6 (50) | 8 (47)
Dizziness (Nervous system disorders) | 2 (2) | 4 (7) | 3 (4) | 2 (5)
Paraesthesia (Nervous system disorders) | 2 (6) | 0 (0) | 2 (3) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (8) | 0 (0) | 1 (20)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (8) | 2 (2) | 4 (16) | 2 (3)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6) | 12 (17) | 4 (5)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (4) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 5 (6) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Acne cystic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (3)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 13 (13) | 8 (9)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (14)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (7) | 3 (5) | 5 (6) | 9 (14)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 2 (3) | 4 (4) | 3 (24)
Abscess rupture (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 2 (3)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 3 (4) | 3 (3) | 1 (2)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (13)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 4 (5) | 2 (3) | 3 (7)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vulvitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 5 (6) | 5 (8) | 2 (8)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 3 (7) | 5 (6) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (2) | 2 (3) | 0 (0) | 2 (13)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (7)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 10 (32) | 10 (34) | 5 (45)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Medical device site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (7) | 5 (8) | 7 (8)
Swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (6)
Contusion (Injury, poisoning and procedural complications) | 3 (11) | 0 (0) | 3 (5) | 2 (2)
Extraskeletal ossification (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 6 (11) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular access site swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (5) | 0 (0) | 1 (3) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Crystal urine present (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sebaceous naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Perineal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03188666/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03188666/SAP_001.pdf